CLINICAL TRIAL: NCT01691807
Title: An Open-label Phase I Drug-drug Interaction Study of Ofatumumab With Bendamustine for the Treatment of Subjects With Indolent B-cell Non-Hodgkin's Lymphoma
Brief Title: Drug-drug Interaction Study of Ofatumumab With Bendamustine in Subjects With Indolent B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113603
Record Dates: First submitted 2012-09-13; First posted 2012-09-25 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Cancer
Keywords: Non-Hodgkin's Lymphoma; drug-drug interaction; ofatumumab; bendamustine
MeSH Terms: conditions — Neoplasms; Lymphoma, Non-Hodgkin | interventions — ofatumumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): bendamustine and ofatumumab treatment of NHL
  Interventions: Drug: ofatumumab; Drug: bendamustine
- Arm B (Experimental): ofatumumab only treatment of NHL
  Interventions: Drug: ofatumumab

INTERVENTIONS:
Drug: ofatumumab — treatment for NHL
Drug: bendamustine — treatment for NHL
  Arms: Arm A

SUMMARY:
The purpose of this study is to evaluate the potential drug-drug interactions between ofatumumab and bendamustine in subjects with previously untreated or relapsed indolent B-cell non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the potential drug-drug interactions between ofatumumab and bendamustine in subjects with previously untreated or relapsed indolent B-cell non-Hodgkin's lymphoma (NHL). Ofatumumab and bendamustine will be administered alone and in combination in a two-arm, open-label study to evaluate the pharmacokinetic profile, safety, tolerability, and efficacy of ofatumumab and bendamustine.

The primary objective of the study is to evaluate pharmacokinetic parameters of ofatumumab and bendamustine alone and in combination. Secondary objectives are to evaluate safety, tolerability, and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with previously untreated or relapsed indolent B-cell NHL requiring treatment. Indolent NHL is defined as small lymphocytic lymphoma (SLL), lymphoplasmacytic lymphoma (LPL), marginal zone lymphoma (MZL), and follicular lymphoma (FL); grades 1, 2, and 3A, defined according to WHO guidelines. Tumor verified to be CD20+ positive from a previous or current lymph node biopsy.
* At least 4 weeks after previous anti-cancer chemotherapy, or radiotherapy treatment.
* At least 12 weeks after previous anti-CD20 radioimmunotherapy, anti-CD20 antibody treatment, and non-anti-CD20 monoclonal antibody treatment.
* Subjects who give consent to this study participation and sign the informed consent form.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
* Age greater than or equal to 18 years at informed consent.
* A female subject is eligible to participate if she is of Non-childbearing potential or required to use a contraception method.
* Male subjects with female partners of child-bearing potential must agree to use a contraception method.
* Subjects must agree to use contraception until 12 months after the last dose of study drug.

Exclusion Criteria:

* Subjects who failed to achieve a complete remission (CR) or partial remission (PR) or progressed within 6 months of last rituximab-containing therapy
* Previous treatment with ofatumumab.
* Prior bendamustine treatment not resulting in a complete remission and partial remission for at least 6 months.
* Previous allogeneic stem cell transplant.
* Previous autologous stem cell transplant.
* High dose steroids greater than or equal to 100 mg prednisone/day (or equivalent) for greater than or equal to 7 consecutive days, given as concomitant medication, within 3 months prior to randomization. No more than 20 mg prednisone or equivalent daily at the time of randomization.
* Grade 3b follicular lymphoma or evidence that the indolent lymphoma has transformed to aggressive lymphoma as verified by biopsy confirmation.
* Known central nervous system involvement by NHL.
* Other past or current malignancy. Subjects who have been free of malignancy for at least 2 years, or have a history of definitively treated non-melanoma skin cancer, or successfully treated in situ carcinoma, are eligible.
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis, and active Hepatitis B or C. Prophylactic antibiotics to prevent recurrent of a prior infection (such as shingles, sinusitis or upper respiratory infection) is allowed.
* Clinically significant cardiac disease as judged by the investigator, including unstable angina, acute myocardial infarction within 6 months of randomization, and uncontrolled congestive heart failure (CHF) or arrhythmia. Patients with a history of CHF or arrhythmia are eligible if their cardiac disease is well controlled on a stable medical regimen.
* History of significant cerebrovascular disease or event with significant symptoms or sequelae (as judged by the investigator).
* Significant concurrent, uncontrolled medical condition that in the opinion of the investigator contraindicates participation this study.
* Positive serology for Hepatitis B (HB) defined as a positive test for Hepatitis B surface antigen (HBsAg). In addition, if negative for HBsAg but Hepatitis B core antibody (HBcAb) positive (regardless of Hepatitis B surface antibody [HBsAb] status), a HB DNA test will be performed and if positive the subject will be excluded. If HBV DNA is negative, the subject may be included but must undergo Hepatitis B virus (HBV) DNA monitoring (see Section 7.7.5). Prophylactic antiviral therapy may be initiated at the discretion of the investigator.
* Current active liver or biliary disease (subjects with Gilbert's syndrome or asymptomatic gallstones, liver metastases related to indolent NHL or otherwise stable chronic liver disease per investigator assessment, are eligible).
* Known human immunodeficiency virus (HIV) positive.
* Screening laboratory values:

  * platelets < 100 x 109/L (unless due to lymphoma involvement of the bone marrow)
  * neutrophils < 1.5 x 109/L (unless due to lymphoma involvement of the bone marrow)
  * serum creatinine > 1.5 times the institution's upper limit of normal (ULN); subjects with a serum creatinine > 1.5 ULN will be eligible if the calculated creatinine clearance [Cockcroft, 1976] or creatinine clearance from a 24-hour urine collection is ≥ 40 mL/min
  * total bilirubin > 1.5 times ULN (unless due to liver involvement by lymphoma or Gilbert's syndrome)
  * transaminases > 2 times ULN
* Known or suspected hypersensitivity to ofatumumab, bendamustine, or mannitol.
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half-lives or 4 weeks prior to Visit 1, whichever is longer or currently participating in any other interventional clinical study
* Lactating women, women with a positive pregnancy test at Visit 1, or women (of childbearing potential) as well as men with partners of childbearing potential, who are not willing to use adequate contraception until 12 months after the last dose of study drug. Adequate contraception is defined in Section 8.1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic measures of Cmax and Area Under the Curve by analysis of blood samples for the amount of each drug present at different timepoints. | 4 months
  The amount of ofatumumab and bendamustine in the blood will be measured when given individually or together to obtain Cmax and Area Under the Curve. Bendamustine levels will be collected at Cycles 1 and 2: Predose, 0.25, 0.5, 0.75, 1 (end of infusion), 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, and 24 hours. Ofatumumab will be collected at Cycle 4: Predose, end of infusion, then 1, 2, 24, and 72 hours after end of infusion, then once each on Days 8, 15, and 22.

SECONDARY OUTCOMES:
Changes in vital signs and the number adverse events | 14 months
  Changes in vital signs will be measured during the entire study to determine any effect on the subjects health. Also the recording of all adverse events that occur during the study will be collected for analysis.
Measure the extent of the disease by CT scan or flow cytometry analysis | 14 months
  Dimension measurement assessments by CT scan of disease will be collected at Screen, Cycle 5, 3 month follow up visit, and 6 month follow up visit. Flow cytometry measurements will be collected at Screen and Weeks 1, 2, 5, 13, 21, 41, and 53.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Southaven, Mississippi
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Morgantown, West Virginia